CLINICAL TRIAL: NCT05217355
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center, Phase II Study to Evaluate the Efficacy and Safety of MBA-P01 in Subjects With Moderate to Severe Glabellar Lines
Brief Title: A Phase II Study to Evaluate the Efficacy and Safety of MBA-P01 in Subjects With Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medytox Korea (Industry)
Responsible Party: Sponsor
Organization: Medy-Tox (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT14-KR21GBL201
Record Dates: First submitted 2021-11-29; First posted 2022-02-01 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBA-P01 (Experimental): Experimental group, Dose: 20U
  Interventions: Drug: MBA-P01 (Botulinum toxin A)
- Placebo (Placebo Comparator): Placebo gorup, Normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MBA-P01 (Botulinum toxin A) — MBA-P01 will be injected into the Glabellar line
  Arms: MBA-P01
Drug: Placebo — Placebo will be injected into the Glabellar line
  Arms: Placebo

SUMMARY:
This study is intended to evaluate the efficacy and safety of MBA-P01 compared to placebo in treatment of glabellar lines.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 19 and 65
* Patients attaining ≥grade 2 (moderate) in the investigator's rating of the severity of glabella lines at maximum frown
* Patients who voluntarily sign the informed consent

Exclusion Criteria:

* Patients with the history of facial nerve paralysis
* Patients with the symptoms of eyelid ptosis determined by the investigator
* Marked facial asymmetry, dermatochalasis, deep dermal scarring in the glabellar area, excessively thick sebaceous skin, or the inability to substantially lessen glabellar lines even by physically spreading them apart, as determined by the investigator
* Active skin disease or infection in the treatment area
* History of surgery which may habe altered the anatomy of the corrugator supercilia muscle or the procerus muscle or related nerve
* Prior treatment with permanent filers, synthetic implantation, and/or autologous fat transplantation in the treatment area
* Subject who received the following drugs within 4 weeks prior to the screening

  1. muscle relaxant: Peripherally acting relaxants, Centrally acting muscle relaxants, skeletal muscle relaxants
  2. benzodiazepine: Diazepam, Chlodiazepoxide, Medazepam, Oxazepam, Potassium clorazepate, Lorazepam etc.

     * Subject who takes Muscle relaxants and benzodiazepine stably for 4 weeks can participate the study
* Subject who reveived any of the below facial aesthetic treatments that, in the investigator's opinion, could interfere the evaluation of efficacy

  1. Prior treatment with fillers in the treatment area within 1 year prior to screening (CaHA, Hyaluronic acid, PLLA, PCL etc.)
  2. Facial resurfacing or skin tightening procedure with lase, light or radiofrequency-based system; or any medium depth or deep depth facial chemical peels in the upper face within 6 months prior to screening
* Subject who received Retinois following period

  1. Systemic drug delivery : within 6 months prior to the screening
  2. Local drug delivery : within 3 months prior to the screening
* Patients with medical conditions who may be at greater risk due to the administration of the investigational drugs (e.g.. diseases that may affect the neuromuscular action including Myasthenia Gravis, Lambert-Eaton Syndrome, Amyotrophic Lateral Sclerosis and motor neuropathy)
* Known immunization or hypersensitivity to any botulinum toxin preparations
* Subject who had botulinum toxin treatment within 6 months prior to the screening or planning to receive botulinum toxic treatment during the study period other than study treatment
* Female subjects who are pregnant or nursing, or planning a pregnancy during the study and female subjects of childbearing potential who are not willing to use acceptable form of sontraception
* Subject who are participating in other interventional clinical study or have participated in such a study within 30 dyas prior to screening
* Subjects who are not eligible for this study at the discretion of the investigator

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Facial Wrinkle Scale(FWS) change | 4 weeks
  Proportion of subjects achieving at least a 2-grade decrease from baseline in score of Facial Wrinkle Scale (FWS) (0:none to 3: severe) of Glabellar line at maximum frown

SECONDARY OUTCOMES:
Investigator-rated improvement rate of glabellar lines at maximum frown | Week 8, 12, 16
  The investigator and participant evaluate the participant's GL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe.
Investigator-rated improvement rate of glabellar lines at rest | Week 4, 8, 12, 16
  The investigator and participant evaluate the participant's GL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe.
Participant-rated improvement rate of glabellar lines at maximum frown | Week 4, 8, 12, 16
  The investigator and participant evaluate the participant's GL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe.
Participant-rated improvement rate of glabellar lines at rest | Week 4, 8, 12, 16
  The investigator and participant evaluate the participant's GL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe.
Participant-rated satisfaction after treatment | Week 4, 8, 12, 16
  Proportion of subject achieving at least 5 score in Participant-rated satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-And Univ. Hospital, Seoul, Dongjak-gu, South Korea